CLINICAL TRIAL: NCT06232005
Title: Intralesional Injection of Mitomycin C Following Visual Internal Urethrotomy for Recurrent Urethral Stricture
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS 604/2022
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Urethral Stricture
Keywords: Mitomycin C - Visual Internal Urethrotomy - Urethral Stricture
MeSH Terms: conditions — Urethral Stricture | interventions — Mitomycin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25 Patients with recurrent urethral stricture undergoing visual internal urethrotomy only. (Active Comparator): Standard procedure of visual internal urethrotomy only for urethral stricture
  Interventions: Drug: Mitomycin c
- 25 Patients with recurrent urethral stricture undergoing visual internal urethrotomy with intralesio (Experimental): intralesional injection of mitomycin-c following the standard visual internal urethrotomy
  Interventions: Drug: Mitomycin c

INTERVENTIONS:
Drug: Mitomycin c — injection of antifibrotic drugs in urethral strictures after internal urethrotomy

SUMMARY:
To evaluate the effectiveness of administering mitomycin C through intralesional injection after performing visual internal urethrotomy (VIU) for the treatment of recurring urethral stricture.

DETAILED DESCRIPTION:
Numerous studies have investigated the impact of intralesional administration of antifibrotic drugs on urethral strictures following visual internal urethrotomy (VIU). These drugs include mitomycin C, botulinum toxin A, somatostatin analog, and glucocorticoids. Mitomycin C (MMC) is known for its potent chemotherapeutic and antibiotic properties. It effectively hinders mitosis and fibroblast proliferation, playing a crucial role in tissue healing and scar formation by reducing the release of matrix proteins through the inhibition of proliferative fibroblasts. With its anti-proliferative and anti-scarring characteristics, MMC proves to be a suitable option for treating recurrent urethral strictures.

thus we conduct a randomized controlled trial to evaluate the safety and efficacy of Mitomycin in decrease urethral stricture recurrence.

ELIGIBILITY:
Inclusion Criteria:

* All adult male patients aged above 18 years with a single bulbar urethral stricture measuring less than ( 1.5 cm), and had failed at least one prior intervention for urethral stricture(urethral dilation & VIU) were included in our study

Exclusion Criteria:

* Patients with urethral strictures more than (1.5 cm), multiple urethral strictures, complex stricture, complicated by a fistula or abscess, completely occluded urethral strictures and previous urethroplasty were excluded

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — surgery in male urethra
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Urethral stricture recurrence | 1 year
  is defined as recurrence of LUTS during follow-up visits starting at 3 months till 12 months with difficulty of passing urine and confirmed by a voiding cystourethrogram.

SECONDARY OUTCOMES:
urinary tract infection | 1 month
  post operative complication confirmed by urine culture
uroflowmetery | 1 year
  evaluate of the urine flow during the follow up period

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
I have to gain consent first from the department and the authors of the study